CLINICAL TRIAL: NCT04069858
Title: Maintaining Antiviral Efficacy After Switching to Generic Entecavir, Baracle® in Patients Taking Baraclude® 1 mg for Antiviral Resistant Chronic Hepatitis B; A Noninferiority Study Assessing Non-detection Rate of Hepatitis B Virus DNA
Brief Title: Maintaining Antiviral Efficacy After Switching to Generic Entecavir 1 mg for Chronic Hepatitis B
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Hyung Joon Yim, Professor, Korea University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2106AS0033
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: CHB patients receiving treatment with Baraclude® 1 mg alone or in combination with other nucleos(t)ide analogues for 12 months or longer after the development of antiviral resistance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baracle (Experimental): Chronic hepatitis B patients who swiched to Baracle® 1 mg from Baraclude® 1 mg treatment as mono- or combination therapy after the development of antiviral resistance to nucleos(t)ide analogues
  Interventions: Drug: Switching to Generic Entecavir (Baracle®)

INTERVENTIONS:
Drug: Switching to Generic Entecavir (Baracle®) — switching to Baracle® 1 mg (generic drug) in chronic hepatitis B patients taking Baraclude® 1 mg (brand drug)
  Other Names: Antiviral therapy

SUMMARY:
Entecavir 1 mg is commonly used in patients with chronic hepatitis B (CHB) patients with previous antiviral resistance. This study evaluates the efficacy and safety of switching to generic entecavir 1 mg (Baracle®, Dong-A Science Technology) in CHB patients taking brand name entecavir 1 mg (Baraclude®, Bristol-Myers Squibb) alone or in combination with other nucleos(t)ide analogues after the development of antiviral resistance.

The primary aim is virological response (<20 IU/mL) at 12 months

DETAILED DESCRIPTION:
This study is a prospective single-arm open-label trial. The primary endpoint is virological response (<20 IU/mL) at 12 months after switching treatment.

Patients who satisfy the inclusion and exclusion criteria will switch from Baraclude® 1 mg to Baracle®. Assessment of treatment response at 12 months is performed by comparing undetectable HBV DNA rates between baseline and 12 months after switching therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >19 years old CHB patients
* Confirmed antiviral resistance
* Taking brand entecavir 1 mg for more than 1 year
* HBV DNA < 20 IU/mL
* Compensated liver cirrhosis
* Willing to participate

Exclusion Criteria:

* Failure to meet the inclusion criteria
* Cr>1.5 mg/dL
* Postive HCV Ab
* Decompensated cirrhosis
* Pregnant women
* HCC
* Alcoholics

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-detection rate of hepatitis B virus DNA | 12 months
  undetectable HBV DNA (<20 IU/mL) at 12 months after switching treatment.

SECONDARY OUTCOMES:
Normalization of liver enzyme | 12 months
  ALT < 40 IU/L
Loss of serological markers of hepatitis B e antigen | 12 months
  Loss of HBeAg
Signs of newly developing antiviral resistance | 12 months
  Elevation of hepatitis B virus DNA by 10 fold assessed by real time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Joon Yim, MD, Principal Investigator — Korea University
Locations (1):
- Korea University Ansan Hospital, Ansan, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Background] Korean Association for the Study of the Liver (KASL). KASL clinical practice guidelines for management of chronic hepatitis B. Clin Mol Hepatol. 2019 Jun;25(2):93-159. doi: 10.3350/cmh.2019.1002. Epub 2019 Jun 12. No abstract available. PMID 31185710